CLINICAL TRIAL: NCT05385159
Title: INNOVATIVE TREATMENT OF SCARRED VOCAL FOLDS BY LOCAL INJECTION OF AUTOLOGOUS ADIPOSE-DERIVED STROMAL VASCULAR FRACTION: EFFICACY VERSUS PLACEBO
Acronym: CELLCORDES2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-53; 2020-004227-17 (EudraCT Number)
Record Dates: First submitted 2021-06-09; First posted 2022-05-23 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-10

CONDITIONS: Scarred Vocal Folds

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADSVF group (Experimental): Adults with Scarred vocal folds, congenital (sulcus) or after phonosurgery
  Interventions: Drug: AUTOLOGOUS ADIPOSE-DERIVED STROMAL VASCULAR FRACTION
- Placebo group (Placebo Comparator): Adults with Scarred vocal folds, congenital (sulcus) or after phonosurgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AUTOLOGOUS ADIPOSE-DERIVED STROMAL VASCULAR FRACTION — Adipose tissue removal, ADSVF production and injection of ADSVF will be done on the same day during a short hospital stay
  Arms: ADSVF group
Drug: Placebo — Adipose tissue removal, ADSVF production, cryopreservation of ADSVF and injection of placebo will be done on the same day during a short hospital stay.
  Arms: Placebo group

SUMMARY:
Vocal Folds scarring (whether congenitally or following phonosurgery) can result in a range of symptoms depending on severity and extent, such as hoarseness, breathy voice, increased effort to speak, and voice fatigue. The inability to phonate normally causes both physical and psychological disability, especially for professional communicators (teachers, tradesmen, singers, etc.). There are several therapies currently available but these are often disappointing, as the great complexity of vocal fold microstructure hinders the development of effective therapy. Thus, identification of innovative strategies able to improve vibrational mechanical properties of vocal folds remains an important clinical challenge.

Autologous Adipose-Derived Stromal Vascular Fraction (ADSVF) is recognized as an easily accessible source of cells displaying angiogenic, anti-inflammatory, immunomodulatory and regenerative properties. Recent experimental and clinical reports also supported the anti-fibrotic potential of ADVSF, mainly attributed to the mesenchymal stem/stromal cell subset.

Safety in humans has already been confirmed in several studies, including our previous clinical trial (ClinicalTrials.gov NCT0262246; EudraCT number: 2015-000238-31). The main objective of this phase I/II trial was to measure for the first time the safety and tolerability of autologous ADSVF local injections in patients with scarred vocal folds. No severe adverse events occurred: only some minor adverse events were reported. Moreover, Voice Handicap Index was improved in all patients with a mean improvement from baseline of 40.1/120 and seven patients were considered as responders, defined as an improvement ≥ 18 points.

Based on these observations, we hypothesized that the injection of autologous ADSVF could reduce the process of fibrosis, improve vibration and then dysphonia and quality of life in patients with scarred vocal folds.

In the absence of a reference treatment, the effectiveness of the ADSVF will be compared to a placebo: the local injection of excipients solution.

This study will test efficacy of the autologous ADSVF to treat vocal folds scarring. It is a randomized, double-blind, phase II clinical trial conducted according to a 2-treatment parallel design, with medico-surgical and scientific collaboration.

Recruitment and follow-up of patients will be done in 4 university hospitals by the respective ENT teams (Marseille, Toulouse, Nice and Montpellier): 36 patients will be recruited and treated on a 24 months period.

At inclusion, 36 patients will be randomized (1:1 ratio) into two groups: ADSVF group and placebo group. Adipose tissue removal, ADSVF production and injection of ADSVF or placebo will be done on the same day during a short hospital stay. Patients will be followed and evaluated at 1 and 6 months with self-evaluation (Voice Handicap Index and a 10 points scale), video-laryngo-stroboscopic examination, vocal assessment with perceptive, acoustic and aerodynamic parameters and evaluation of adverse events. At the end of this 6-month follow-up (primary endpoint), patients of each group having tolerated the first injection well but in therapeutic failure (improvement of VHI <18 as described by Jacobson in 1997 or improvement of VHI ≥ 18 but not normal which means > 20 according to Woisard, 2004) will be offered an injection of thawed and washed ADSVF. Patients will continue to be followed in open-label on the same endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Subscription to the French Social Security System
* signed informed consent;
* voice Handicap Index > 50/120;
* scarred vocal folds, congenital (sulcus) or after phonosurgery;
* scarred middle third in videolaryngostroboscopy;
* at least six-months delay after initial surgery if appropriate;
* patients aged between 18 and 70;
* good general condition;
* negative pregnancy test & contraception for women of child-bearing age.

Exclusion Criteria:

* Refusal of speech therapy;
* history of malignant lesion or severe dysplasia of the scarred vocal fold;
* history of laryngeal papillomatosis;
* contraindication to local anesthesia;
* anti-coagulant treatment;
* coagulation disorders (Prothrombin Ratio <65%, Activated Partial Thromboplastin Time >1,2);
* active infectious diseases;
* any active viral infection from among the following: HIV, HTLV I and II, VHB, VHC and Syphilis;
* known sensitivity to human serum albumin (HSA);
* necessity of intraoperative prophylactic antibiotics;
* BMI < 18 kg/m2 to insure adequate abdominal or other subcutaneous adipose tissue accessible to lipoharvest.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Self-evaluation with the Voice Handicap Index | 6 months
  The Voice Handicap Index (VHI) is composed of 3 parts (E = emotional subscale, F = functional subscale, P = physical subscale), with lower scores indicating a better voice perception.
  Patients are considered as responders if they achieved the Minimal Clinically Important Difference (MCID) defined by Jacobson as a shift in the total VHI score of at least 18 / 120 (Jacobson, 1997).

SECONDARY OUTCOMES:
Self-evaluation of dysphonia | 6 months
  on a scale from 0 to 10
Aspect of vibration in videolaryngostroboscopy | 6 months
  For each stroboscopic parameter, a four-point grading scale (0 = no deviance, 3 = severe deviance) is used. Analyses will be done by a single jury in Marseille, in a random order and a blind way
The signal to noise ratio | 6months
  reading of a short text and a sustained vowel: quantifies the aperiodic portion of the voice signal (the higher the signal the better)
  .
The vocal range | 6 months
  reading of a short text and a sustained vowel:difference between the maximum frequency and the minimum frequency
The jitter | 6months
  reading of a short text and a sustained vowel:refers to a short-term (cycle-to-cycle) perturbation in the fundamental voice frequency (the lower the better).

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, PACA, France